CLINICAL TRIAL: NCT04296656
Title: Mothers' Parenting Satisfaction and Parenting Self-efficacy During the Postpartum Period: An Evaluation of a Infant Calming Method
Brief Title: Mothers' Parenting Satisfaction and Parenting Self-efficacy: An Evaluation of a Infant Calming Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R18188H
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Parenting Satisfaction; Parenting Self-efficacy
Keywords: parenting satisfaction; parenting self-efficacy; behavioral infant calming intervention

STUDY DESIGN:
Intervention Model Description: Mothers in the intervention group were taught the infant calming intervention (the 5 S's). The mothers in both control and intervention groups received standard care and support provided by the midwives on the postpartum wards. Baseline data were collected before randomization in the hospital. Follow-up data were collected six to eight weeks postpartum at home.
  The research groups were randomized in the following way: The mothers who were on one of the postpartum wards during the days when the intervention (5 S's) were taught, were randomly allocated to the group during the data collection period. The intervention was executed every second week, three days a week on Mondays, Wednesdays and Fridays. The intervention was executed until 120 mothers had participated in them. Control group mothers (n = 130) were recruited by in a similar fashion as the intervention group, but on alternate weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Mothers in the intervention group were taught the infant calming technique 5 S's, a part of The Happiest Baby (THB) method. THB is based on the theory that infants have an innate "calming reflex" that can soothe infant fussing, excessive crying and prolong sleep. This reflex is triggered by five activities that mimic the sensory milieu of the womb. The 5 S's include swaddling, side position, sound (white noise), swing and suck.
  The intervention consisted of a 20-minute face-to-face guidance session with the researcher, executed individually in the mother's hospital room. Each mother was given a leaflet to take home that explained the 5 steps in short. Safety issues, such as safest sleep position (supine), allowing hips to flex and how to avoid overheating when swaddled, were addressed. The same researcher executed each guidance session to maintain standardization.
  Interventions: Behavioral: The 5 S's infant calming intervention
- Control group (No Intervention): Standard care on postpartum ward (breastfeeding and infant care guidance and support in recovering from childbirth and transitioning into parenthood).

INTERVENTIONS:
Behavioral: The 5 S's infant calming intervention — 5 simple steps to calm a fussy or crying infant. Steps include swaddling, side position, sound (white noise), swing and suck.
  Arms: Intervention group

SUMMARY:
The main aim of this study is to investigate how to support families with an excessively crying or fussy infant during the first months of the child. The purpose is to discover how an excessively crying or fussy infant affects the mothers' parenting satisfaction and parenting self-efficacy. Furthermore the purpose is to investigate how a behavioral intervention (The 5 S's) affects the infants' mothers' parenting satisfaction and self-efficacy and to evaluate the effectiveness of the intervention.

DETAILED DESCRIPTION:
This is a randomized controlled follow-up parallel trial that compares PSE and PS in an intervention and control group. The data was collected during March 1st to May 20th, 2019 from three postpartum wards. The mothers were recruited by midwives on the wards after childbirth. The baseline sample size was 250 mothers, which is based on a conducted power analysis. The sample size calculation was based on previous study, from which the standard deviation (0.81) for change in parental satisfaction was calculated. Baseline data were collected before randomization in the hospital. Follow-up data were collected six to eight weeks postpartum at home.

The instruments to assess the study outcomes were the parenting self-efficacy (PSE) scale developed and validated by Salonen et al. and parenting satisfaction (PS) scale, the evaluation subscale of the questionnaire "What Being the Parent of a New Baby is Like" by Pridham & Chang, 1989.

Data were analyzed with SPSS statistical software for Windows, release 25. Descriptive statistics included frequencies, percentages, means and medians. Total scores for the PSE instrument and WBPL-R evaluation subscale (PS) were calculated by summing the scores for all items and dividing the sum by the number of items. Higher scores indicated better outcomes. Comparisons between groups were made of mother characteristics, PSE and PS. Due to skewed distributions, non-parametric tests were used. Mann-Whitney U tests were used for two group comparisons, and Kruskal Wallis tests were used for three or more group comparisons.

Results have not yet been reported.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous mothers
* Multiparous mothers
* Mothers of healthy infants rooming in (with mother)

Exclusion Criteria:

* Mothers with infants who were treated on another ward during data collection
* Mothers with multiple infants
* Mothers with inability to understand Finnish

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Parenting satisfaction (PS) | Baseline
  The questionnaire "What Being the Parent of a New Baby is Like" measures parenting satisfaction and has three distinct subscales: evaluation (11 items), centrality (8 items), and life change (6 items). The Evaluation subscale contains 11 items where the mothers responded on a nine-point scale with verbal end anchors, such as 1 = not at all (satisfied) to 9 = completely (satisfied). Higher scores indicate more PS. The evaluation subscale contains items such as "How well do you know your baby?", "How satisfied are you in being a parent of a new baby?" and "How satisfied are you with baby care tasks?".
Change in Parenting satisfaction (PS) | 6-8 weeks postpartum
  The questionnaire "What Being the Parent of a New Baby is Like" measures parenting satisfaction and has three distinct subscales: evaluation (11 items), centrality (8 items), and life change (6 items). The Evaluation subscale contains 11 items where the mothers responded on a nine-point scale with verbal end anchors, such as 1 = not at all (satisfied) to 9 = completely (satisfied). Higher scores indicate more PS. The evaluation subscale contains items such as "How well do you know your baby?", "How satisfied are you in being a parent of a new baby?" and "How satisfied are you with baby care tasks?".
Parenting Self-Efficacy (PSE) | Baseline
  This questionnaire measures parenting self efficacy and is domain-specific, and it includes 27 items measuring different infant care skills. These skills are cognitive skills (11 items) such as "I know how to calm a crying baby", affective skills (seven items) such as "I know what my baby enjoys" and behavioural skills (nine items) such as "I'm able to put my baby to sleep". The instrument has a six-point Likert scale 1 = "strongly disagree" to 6 = "strongly agree". Total parenting self-efficacy scores were calculated by adding up the scores of all items and dividing the sum by the number of items. In addition, the score for each subcategory was calculated by adding up the scores of all items in the subcategory and dividing the sum by the number of items. In this instrument, higher scores indicate better outcomes.
Change in Parenting Self-Efficacy (PSE) | 6-8 weeks postpartum
  This questionnaire measures parenting self efficacy and is domain-specific, and it includes 27 items measuring different infant care skills. These skills are cognitive skills (11 items) such as "I know how to calm a crying baby", affective skills (seven items) such as "I know what my baby enjoys" and behavioural skills (nine items) such as "I'm able to put my baby to sleep". The instrument has a six-point Likert scale 1 = "strongly disagree" to 6 = "strongly agree". Total parenting self-efficacy scores were calculated by adding up the scores of all items and dividing the sum by the number of items. In addition, the score for each subcategory was calculated by adding up the scores of all items in the subcategory and dividing the sum by the number of items. In this instrument, higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication, also Study Protocol will be allowed in 2022, after discussions and in good cooperation with Tampere University Hospital.
Supporting Information: Study Protocol, CSR
Time Frame: 2022-2027
Access Criteria: Permission from Tampere University Hospital